CLINICAL TRIAL: NCT00845598
Title: A Proof of Concept Study to Evaluate Comparative Efficacy of an Azelastine/Fluticasone Combination Nasal Spray vs. Twice the Dose of Fluticasone in Persistent Allergic Rhinitis
Brief Title: Azelastine Fluticasone Combination vs. Fluticasone
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Could not get IMP
Sponsor: University of Dundee (Other)
Responsible Party: Principal Investigator, Brian J Lipworth, Professor, University of Dundee
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: VAI04
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Allergic Rhinitis
Keywords: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — azelastine; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azelastine Fluticasone (Experimental)
  Interventions: Drug: Azelastine , fluticasone
- Fluticasone propionate (Active Comparator)
  Interventions: Drug: Fluticasone propionate

INTERVENTIONS:
Drug: Azelastine , fluticasone — Azelastine Hydrochloride BP 0.10% w/v AND Fluticasone propionate BP 0.0357% w/v as combination
  1 squirt in each nostril twice daily
  Arms: Azelastine Fluticasone
Drug: Fluticasone propionate — Fluticasone propionate 0.05% w/w 2 squirts in each nostril (50 μg per squirt)
  Arms: Fluticasone propionate

SUMMARY:
The purpose of this study is to see how a combination spray of azelastine and fluticasone (antihistamine and steroid) compares with a steroid nasal spray (fluticasone) alone in allergic rhinitis i.e. does azelastine permit the use of lesser steroid dose (steroid sparing effect) to achieve the same benefit.

DETAILED DESCRIPTION:
Allergic rhinitis (AR) is a major chronic respiratory disease with a prevalence approaching nearly 25% in the worldwide population.Allergic Rhinitis is a common and relatively undiagnosed public health problem and has been reported as being one of the ten most common causes for outpatient attendances to the general practitioner. Long term untreated allergic rhinitis may lead on to asthma. When exposed to allergens (pollen, house dust mite etc) in the atmosphere, the mast cells in the nose burst and an inflammatory response is triggered and patients experience sneezing, itching, blocked nose and running. These allergens may be used as provocation agents to recreate the disease symptoms to confirm the diagnosis of which allergens one is allergic to. However, there is a risk of allergic reactions in doing so. Adenosine monophosphate (AMP)achieves the same goal by stimulating the mast cells and causing them to burst without actually the risks of allergen provocation tests. Such tests are now commonplace in research and clinical medicine. Nasal steroids are considered to be the most potent medications for allergic rhinitis, particularly nasal blockage. Nasal antihistamines are also available but they act mainly to limit nasal running, itching and sneezing and have lesser effect on blockage. The other advantage is that they act very quickly while steroids take at least 72 hours to begin acting and weeks to achieve maximal benefit. Finally, they are free of significant short and long term side effects. Having said that nasal steroids are very safe and unlike inhaled or oral steroids have not been shown to cause systemic side effects in adults. Therefore, it is interesting to see if a combination of an antihistamine and nasal steroid would add their good qualities mentioned above and by the act of reducing the dose of steroid reduce their side effects. To do this we will use nasal AMP challenge as an outcome measure as we have done research studies for over a decade with. We will look at noninvasive nasal airflow parameters, nasal nitric oxide levels, and for safety we will look at the overnight urinary cortisol and creatinine ratio which is the most sensitive and noninvasive test of urine to quantify how much steroid has been absorbed in the blood stream.

ELIGIBILITY:
Inclusion Criteria:

* Male of Female aged 18-65 years.
* Persistent allergic rhinitis with or without asthma.
* Atopy to at least one allergen on SPT.
* Ability to give a written informed consent.
* Ability and willingness to comply with the requirements of the protocol.

Exclusion Criteria:

* Recent respiratory tract/sinus infection within the last 2 months. .
* Pregnancy, planned pregnancy or lactation.
* Known or suspected hypersensitivity to any of the IMP's.
* Concomitant use of medicines (prescribed, OTC or herbal) like alpha blockers that may interfere with the trial.
* Nasal Polyposis grade 2+, Deviated nasal septum ≥ 50%
* The use of oral corticosteroids within the last 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Maximum percentage fall in PNIF after 400mg/ml of AMP nasal challenge between both groups. | 0, 2 weeks, 4 weeks, 6 weeks, 8 weeks

SECONDARY OUTCOMES:
60 minute recovery to AMP challenge | 0, 2 weeks, 4 weeks, 6 weeks, 8 weeks
Mini RQLQ | 0, 2 weeks, 4 weeks, 6 weeks, 8 weeks
Global visual analogue scale | 0, 2 weeks, 4 weeks, 6 weeks, 8 weeks
Nasal lavage for cytokines | 0, 2 weeks, 4 weeks, 6 weeks, 8 weeks
Overnight urinary cortisol creatinine ratio | 0, 2 weeks, 4 weeks, 6 weeks, 8 weeks
Domiciliary diary cards | 2 week treatment periods

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Vaidyanathan, MBBS, Principal Investigator — University of Dundee; Brian Lipworth, MD, FRCP, Study Director — University of Dundee
Locations (2):
- United Kingdom (2):
  - Ninewells Hospital and Medical School, Dundee
  - Perth Royal Infirmary, Perth

REFERENCES:
- [Background] Bousquet J, Van Cauwenberge P, Khaltaev N; Aria Workshop Group; World Health Organization. Allergic rhinitis and its impact on asthma. J Allergy Clin Immunol. 2001 Nov;108(5 Suppl):S147-334. doi: 10.1067/mai.2001.118891. No abstract available. PMID 11707753
- [Background] Nassef M, Shapiro G, Casale TB; Respiratory and Allergic Disease Foundation. Identifying and managing rhinitis and its subtypes: allergic and nonallergic components--a consensus report and materials from the Respiratory and Allergic Disease Foundation. Curr Med Res Opin. 2006 Dec;22(12):2541-8. doi: 10.1185/030079906x158057. PMID 17265594
- [Background] Nolte H, Nepper-Christensen S, Backer V. Unawareness and undertreatment of asthma and allergic rhinitis in a general population. Respir Med. 2006 Feb;100(2):354-62. doi: 10.1016/j.rmed.2005.05.012. Epub 2005 Jul 11. PMID 16005621
- [Background] Gupta R, Sheikh A, Strachan DP, Anderson HR. Burden of allergic disease in the UK: secondary analyses of national databases. Clin Exp Allergy. 2004 Apr;34(4):520-6. doi: 10.1111/j.1365-2222.2004.1935.x. PMID 15080802
- [Background] Weiner JM, Abramson MJ, Puy RM. Intranasal corticosteroids versus oral H1 receptor antagonists in allergic rhinitis: systematic review of randomised controlled trials. BMJ. 1998 Dec 12;317(7173):1624-9. doi: 10.1136/bmj.317.7173.1624. PMID 9848901
- [Background] Meltzer EO, Weiler JM, Dockhorn RJ, Widlitz MD, Freitag JJ. Azelastine nasal spray in the management of seasonal allergic rhinitis. Ann Allergy. 1994 Apr;72(4):354-9. PMID 7908778
- [Background] Newson-Smith G, Powell M, Baehre M, Garnham SP, MacMahon MT. A placebo controlled study comparing the efficacy of intranasal azelastine and beclomethasone in the treatment of seasonal allergic rhinitis. Eur Arch Otorhinolaryngol. 1997;254(5):236-41. doi: 10.1007/BF00874095. PMID 9195148
- [Background] Berger WE, Fineman SM, Lieberman P, Miles RM. Double-blind trials of azelastine nasal spray monotherapy versus combination therapy with loratadine tablets and beclomethasone nasal spray in patients with seasonal allergic rhinitis. Rhinitis Study Groups. Ann Allergy Asthma Immunol. 1999 Jun;82(6):535-41. doi: 10.1016/s1081-1206(10)63161-4. PMID 10400480